CLINICAL TRIAL: NCT00001671
Title: The Nosology and Etiology of Leukodystrophies of Unknown Cause
Brief Title: The Classification and Cause of Leukodystrophies of Unknown Cause
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 970170; 97-N-0170
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2008-12-15

CONDITIONS: Lysosomal Storage Disease
Keywords: White Matter; Myelin; Degenerative Diseases; Genetic; Oligodendrocytes; Leukodystrophy
MeSH Terms: conditions — Lysosomal Storage Diseases

SUMMARY:
Leukodystrophy is a disease of the white matter of the brain. White matter is the portion of the brain responsible for conducting electrical impulses from one area of the brain to the other. Insulating cells called myelin cover the brain and nerve cells in the white matter. If myelin becomes damaged electrical information cannot be transferred properly.

Many patients suffering from leukodystrophies do not fit the description of any of the defined types of leukodystrophies and are therefore considered to have a leukodystrophy of unknown cause.

The purpose of this study is to define groups of patients with leukodystrophies and to work toward finding the cause of the disorders. In order to do this, researchers will analyze patients with leukodystrophies of unknown causes. Patients will undergo clinical, neurophysiologic, biochemical, and genetic examinations and tests.

Researchers believe that by studying these patients and their disorders they will be able to better understand the causes of myelin destruction, and eventually lead to effective treatments for these disorders.

DETAILED DESCRIPTION:
Patients with leukodystrophies (LDs) of unknown etiology are a heterogeneous group but constitute the second largest group of genetic white matter diseases. The purpose of this study is to: (a) define novel homogeneous groups of patients with LDs and (b) work toward finding the cause of these disorders. In order to achieve these goals, patients with LDs of unknown cause will be analyzed clinically, neurophysiologically, biochemically and genetically. Patients would have been diagnosed as having no known leukodystrophies at outside centers. At the Clinical Center, such patients will undergo a series of neuropsychological, blood, urine, spinal fluid, radiological, and peripheral tissue pathological tests. Some of these tests will be part of a standard battery while others will be tailored to individual patients. Patients will be followed for 3 years. Patients will be screened for mutations in genes coding for structural myelin proteins. In some patients in whom all tests yielded no information regarding the etiology of their disease, open brain biopsy will be considered. Brain biopsy tissue will be evaluated using a novel combination of approaches including detailed pathological, immunohistochemical, and biochemical analysis of myelin proteins and lipids. Oligodendroglial biology and expression of myelin genes in the brain will also be investigated in situ. It is hoped that the present study will help clarify the nosology of the leukodystrophies and significantly advance our understanding of the pathogenesis of these diseases.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Candidates for participation in the protocol will be patients of all ages with clinical and radiographic signs of leukodystrophy who do not have a specific etiology despite a previous comprehensive workup. The preceding investigation would have excluded the following: adrenoleukodystrophy, adrenomyeloneuropathy, metachromatic leukodystrophy, Krabbe disease, Canavan disease, a well-defined amino acid organic acid disorder, or a systemic mitochondrial cytopathy.
  2. First -degree relatives of patients with leukodystrophies of unknown etiology (father, mother, siblings, or sons and daughters of the patients)

EXCLUSION CRITERIA:

1. Refusal to sign the protocol consent form.
2. Candidates who are unable to travel to the National Institutes of Health Clinical Center.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400
Dates: Start 1997-09-09; Study Completion 2008-12-15

CONTACTS AND LOCATIONS:
Locations (5):
- United States (2):
  - University of California, San Francisco, San Francisco, California
  - Childrens National Medical Center, Washington D.C., District of Columbia
- Institut National de la Sante' et de la Recherche Medicale, Clermont-Ferrand, Cedex, France
- Tel Aviv University, Tel Aviv, Israel
- Academiseh Ziuekenhuis Vrije Universiteit, Amsterdam, Netherlands

REFERENCES:
- [Background] Aicardi J. The inherited leukodystrophies: a clinical overview. J Inherit Metab Dis. 1993;16(4):733-43. doi: 10.1007/BF00711905. PMID 7692130
- [Background] Schiffmann R, Moller JR, Trapp BD, Shih HH, Farrer RG, Katz DA, Alger JR, Parker CC, Hauer PE, Kaneski CR, et al. Childhood ataxia with diffuse central nervous system hypomyelination. Ann Neurol. 1994 Mar;35(3):331-40. doi: 10.1002/ana.410350314. PMID 8122885
- [Background] Schiffmann R, Tedeschi G, Kinkel RP, Trapp BD, Frank JA, Kaneski CR, Brady RO, Barton NW, Nelson L, Yanovski JA. Leukodystrophy in patients with ovarian dysgenesis. Ann Neurol. 1997 May;41(5):654-61. doi: 10.1002/ana.410410515. PMID 9153528
- [Derived] McNeill N, Nasca A, Reyes A, Lemoine B, Cantarel B, Vanderver A, Schiffmann R, Ghezzi D. Functionally pathogenic EARS2 variants in vitro may not manifest a phenotype in vivo. Neurol Genet. 2017 Jul 14;3(4):e162. doi: 10.1212/NXG.0000000000000162. eCollection 2017 Aug. PMID 28748214